CLINICAL TRIAL: NCT05281289
Title: Effect of Kinesio Tape Application and Stretching Exercises on Calf Cramps During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/003151
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Calf Cramps During Pregnancy
Keywords: kinesio-tape,stretching exercises, calf cramps, pregnants, cramp questionnaire
MeSH Terms: interventions — Athletic Tape; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-tape application+stretchinge exercises (Experimental): the patient received A"Ystrip"of KT was applied to the testing leg 30% tension for 48h and was asked to assume comfortable supine position and the therapist applied 15 seconds of passive stretch to the calf muscle followed by 30 seconds of rest and this exercise was repeated 6 times per session for 2 days and ecieved instructions about dealing with calf cramps with self low sustained stretch of calf muscle.
  Interventions: Other: kinesio-tape; Other: stretching exercise; Other: instructions about dealing with calf cramps
- self low sustained strestch (Experimental): the patient recieved instructions about dealing with calf cramps with self low sustained stretch of calf muscle.
  Interventions: Other: instructions about dealing with calf cramps

INTERVENTIONS:
Other: kinesio-tape — KT is comprised of a polymer elastic strand warped by 100% cotton fibers and designed to allow a longitudinal stretch of 55-60% of its resting length.
  Arms: Kinesio-tape application+stretchinge exercises
Other: stretching exercise — 15 seconds of passive stretching exercise for calf muscle followed by 30 seconds of rest
  Arms: Kinesio-tape application+stretchinge exercises
Other: instructions about dealing with calf cramps — instructions about dealing with calf cramps by self low sustained stretch of calf muscle

SUMMARY:
The aim of this study is to investigate the effect of kinesio-tape application and stretching exercise on calf muscle cramp during pregnancy

DETAILED DESCRIPTION:
Up to 30% to 50% of pregnant women suffered from leg cramps, especially in the third trimester. Almost two-thirds of these women experience leg cramps twice per week and they can occur at any time, particularly at night.In mild and moderate cases, calf cramps may last for seconds, but in severe cases, leg cramps in pregnancy may last for minutes .In many cases calf cramps are very painful , which can affect daily activities, restrict exercise and performance, motive sleep disturbance and reduce the quality of life.Non-drug treatments are found to being effective for the treatment of muscle cramps. Non-drug treatments such as muscle stretching, physical exercise, avoidance of physical fatigue, massage, relaxation, heat therapy, weight loss, sensory nerve stimulation, ankle splints worn while sleeping, and changes to sleeping and sitting positions.This study has two groups; one recieved kinesio-tape application and stretching exercises and the second one recieved instructions about dealing with cramps with self low sustained stretch

ELIGIBILITY:
Inclusion Criteria:

* pregnant women who are suffering from calf cramps.
* Their age range from 25 to 35 years.
* Their body mass index range from 25 to 29.9 kg/m2 .

Exclusion Criteria:

* Skin abnormalities (skin malignancy in the treated area or burned).
* History of previous back surgery.
* Neuromuscular diseases like multiple sclerosis.
* Sensory disturbances.
* Evidence of previous vertebral fractures or major spinal structural abnormality, spondylolisthesis or spinal stenosis.
* Systemic disease of musculoskeletal system.
* Viscerogenic cause of back pain.
* Also, women who have eclampsia or pre-eclampsia.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
calf pain intensity | 2days
  cramp VAS is used to measure pain intensity

SECONDARY OUTCOMES:
weight bearing ankle dorsiflexion ROM | 2days
  weight bearing ankle dorsiflexion ROM is measured by digital inclinometer
straight leg raising ROM | 2days
  straight leg raising ROM is measured by digital inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt